CLINICAL TRIAL: NCT06100692
Title: Effect of Prophylactic Use of Oral Vitamin D and Zinc in Management of the Severity of Radiation Induced Oral Mucositis of Head and Neck Cancer Patients
Brief Title: Prophylactic Oral Vitamin D and Zinc for Radiation-Induced Oral Mucositis in Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shorooq Mostafa Kamel Ahmed, resident doctor at clinical oncology and nuclear medicine, Assiut University
Other Study IDs: EPUO
Record Dates: First submitted 2023-10-14; First posted 2023-10-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Vitamin D; Zinc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vit D and zinc group: will receive combination of oral vit D and zinc 30 patients
  Interventions: Drug: Vitamin D
- placebo group: receive Placebo or no treatment 30 patients

INTERVENTIONS:
Drug: Vitamin D — the patients will receive a 30 pts a combination of oral vit D and zinc
  Other Names: zinc
  Groups: vit D and zinc group

SUMMARY:
The main aim of this study was to evaluate clinically the effect of a combination between oral vitamin D and oral zinc in comparison to conventional therapy in prevention of radiotherapy-induced oral mucositis in Assiut University Hospitals.

DETAILED DESCRIPTION:
Most head and neck cancers are derived from the mucosal epithelium in the oral cavity, pharynx and larynx and are known collectively as head and neck squamous cell carcinoma (HNSCC). Oral cavity and larynx cancers are generally associated with tobacco consumption, alcohol abuse or both, whereas pharynx cancers are increasingly attributed to infection with human papillomavirus (HPV), primarily HPV-16. Thus, HNSCC can be separated into HPV-negative and HPV-positive HNSCC.

As a major histological type of HNC, head and neck squamous cell carcinoma (HNSCC) is the sixth most common cancer worldwide. Totally, 53,000 new cases and 10,860 HNC-related deaths were observed in the U.S. in 2019. According to the estimation of the World Health Organization, 439,000 mouth and oropharynx cancer will be observed in 2030.

The main treatment options are surgery, radiation therapy, chemotherapy, targeted therapy, and immunotherapy.

Treatment options and recommendations depend on several factors, including the type and stage of head and neck cancer, possible side effects, and the patient's preferences and overall health.

Radiation therapy (RT) plays a key role in curative-intent treatments for head and neck cancers. Its use is indicated as a sole therapy in early stage tumors or in combination with surgery or concurrent chemotherapy in advanced stages. Recent technologic advances have resulted in both improved oncologic results and expansion of the indications for RT in clinical practice.

Chemotherapy is a treatment for head and neck cancer that uses powerful drugs to attack cancer cells. Often chemotherapy drugs are given before or during radiation to improve the effectiveness of care. Other drug therapies target the genetic mutations found in tumors or stimulate the immune system to fight the cancer.

Approximately 60% of head and neck cancer patients who were instructed to receive radiotherapy will suffer from oral mucositis. More importantly, the incidence of oral mucositis increases to 90% when patients underwent concurrent chemotherapy 19% of the latter will be hospitalized and will experience a delay in antineoplastic treatment for high-grade mucositis management.

Oral mucositis is a common side-effect associated with systemic chemotherapy and radiation of the head and neck region. It is characterized as an inflammation of the oral mucous membranes accompanied by many complex mucosal and submucosal changes. Ulcerative oral mucositis can cause significant oral pain, impair nutritional intake, lead to local or systemic infection, and cause significant economic cost. In addition, it may necessitate interruptions in cancer therapy, resulting in a reduction of the quality of life, a worse prognosis and an increase in patient management costs, thus adversely affecting patient prognosis.

vitamin D is a fat soluble vitamin which has important calcemic roles in the body regarding bone homeostasis and calcium/phosphorus balance. Recently, the non-calcemic roles of vitamin D as anti-inflammatory, anti-oxidant and immuno-regulatory functions have been widely reported.So, we tried to use it for prevention of radiation induced oral mucositis

Oral mucositis scale Vitamin D supplementation significantly improved erythema, lichenoid, edema, ulceration and pain in patients with inoperable/unresectable oral cancer.

Hypovitaminosis D could increase risk of developing OSCC from OPMDs, thus altering the immune response and it is associated with a lower survival rate in patients with OSCC, a greater recurrence of tumors in patients who underwent surgical treatment, and an increase in adverse reactions to chemotherapy. The use of vitamin D supplements can be a complement to primary therapy to prevent the recurrence of lesions and reduce adverse events associated with treatment.

Vitamin D supplementation has a role in reducing treatment-related toxicities, especially in advanced cancer.

Zinc sulfate is beneficial in decreasing the severity of radiation-induced mucositis and oral discomfort. These results should be confirmed by additional evaluation in randomized studies with a larger number of patients.

zinc has the potential of relieving oxidant damage and the progression of reactive oxygen species (ROS)-induced disease.

The World Health Organization has developed a grading system for mucositis based on clinical appearance and functional status.

The WHO scale is dependent on both objective and subjective variables, and measures anatomical, symptomatic as well as functional components of oral mucositis.

WHO Oral Mucositis Grading Scale Grade Description 0 (none) None I (mild) Oral soreness, erythema II (moderate) Oral erythema, ulcers, solid diet tolerated III (severe) Oral ulcers, liquid diet only IV (life-threatening) Oral alimentation impossible

ELIGIBILITY:
Inclusion Criteria:

* Selection of patients

  1. All adults (18 years or older ), who were confirmed based on pathology ( Head and Neck Squamous Cell Carcinomas ), will administere chemo-radiotherapy either as preoperative (neoadjuvant), postoperative (adjuvant) therapy or definitive therapy, no randomization .
  2. The treatment group will receive combined oral Vit D and Zinc and the control group will take placebo capsules or receive no treatment.
  3. No documentation of any other causes of oral mucositis in their medical records as : immunocomprmized patients d.t HIV

Exclusion Criteria:

1. Non Head and Neck cancer
2. patients with any other causes of oral mucositis
3. Double malignancy
4. Un eligible patients for radiotherapy ( comatosed, bedridden and sever chest disease )

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: maternal and perinatal morbidity and mortality
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
oral mucositis scale | baseline
  The Oral Mucositis Assessment Scale (OMAS) is an objective scale that measures erythema and ulceration at nine sites within the oral cavity grade0:(none) grade1(mild): oral soreness and erythema grade 2(moderate):oral erythema ,ulcers, solid diet tolerance grade 3(sever) :liquids diet only grade 4(life threatening) oral alimentation impossible

REFERENCES:
- [Background] Hashim D, Sartori S, La Vecchia C, Serraino D, Maso LD, Negri E, Smith E, Levi F, Boccia S, Cadoni G, Luu HN, Lee YA, Hashibe M, Boffetta P. Hormone factors play a favorable role in female head and neck cancer risk. Cancer Med. 2017 Aug;6(8):1998-2007. doi: 10.1002/cam4.1136. Epub 2017 Jul 14. PMID 28707400
- [Background] Shuai T, Yi LJ, Tian X, Chen WQ, Chen H, Li XE. Prophylaxis with oral zinc sulfate against radiation-induced oropharyngeal mucositis in patients with head and neck cancer: Protocol for a meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(48):e13310. doi: 10.1097/MD.0000000000013310. PMID 30508920
- [Background] Rambod M, Pasyar N, Ramzi M. The effect of zinc sulfate on prevention, incidence, and severity of mucositis in leukemia patients undergoing chemotherapy. Eur J Oncol Nurs. 2018 Apr;33:14-21. doi: 10.1016/j.ejon.2018.01.007. Epub 2018 Feb 2. PMID 29551172
- [Background] Villa A, Sonis ST. Mucositis: pathobiology and management. Curr Opin Oncol. 2015 May;27(3):159-64. doi: 10.1097/CCO.0000000000000180. PMID 25774860
- [Background] Anand A, Singh S, Sonkar AA, Husain N, Singh KR, Singh S, Kushwaha JK. Expression of vitamin D receptor and vitamin D status in patients with oral neoplasms and effect of vitamin D supplementation on quality of life in advanced cancer treatment. Contemp Oncol (Pozn). 2017;21(2):145-151. doi: 10.5114/wo.2017.68623. Epub 2017 Jun 30. PMID 28947884
- [Background] Sutherland SE, Browman GP. Prophylaxis of oral mucositis in irradiated head-and-neck cancer patients: a proposed classification scheme of interventions and meta-analysis of randomized controlled trials. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):917-30. doi: 10.1016/s0360-3016(00)01456-5. PMID 11240232
- [Background] Pulito C, Cristaudo A, Porta C, Zapperi S, Blandino G, Morrone A, Strano S. Oral mucositis: the hidden side of cancer therapy. J Exp Clin Cancer Res. 2020 Oct 7;39(1):210. doi: 10.1186/s13046-020-01715-7. PMID 33028357